CLINICAL TRIAL: NCT05989425
Title: Surufatinib as Neoadjuvant Treatment for Locally Advanced or Metastatic Differentiated Thyroid Cancer: an Open-label, Multicenter, Single-arm Study
Brief Title: Surufatinib as Neoadjuvant Treatment for Locally Advanced or Metastatic Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chen Jiaying, Professor, Fudan University Shanghai Cancer, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-T102
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surufatinib (Experimental): Surufatinib 300mg will be taken orally once daily continuously through a 28-day cycle of study treatment. After treatment, the patients will receive operation treatment if the tumor is evaluated as resectable cases by clinical examination. Patients with high risk of postoperative recurrence will receive 131I treatment. After 131I treatment, maintenance treatment with surufatinib will be determined according to the recurrence risk stratification.
  Interventions: Drug: surufatinib

INTERVENTIONS:
Drug: surufatinib — Surufatinib is a tablet in the form of 50mg, oral, once a day.

SUMMARY:
Locally advanced thyroid cancer has a wide range of surgery, large trauma and high local recurrence rate. It is one of the main causes of death in patients with thyroid cancer. Therefore, more effective treatments are urgently needed. This study is designed to evaluate the efficacy and safety of the Surufatinib for Locally Advanced Thyroid Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic thyroid cancer confirmed by histology or cytology, including papillary thyroid carcinoma, follicular thyroid carcinoma, poorly differentiated thyroid cancer, particularly differentiated thyroid cancer. Locally advanced stage refers to: 1) Primary tumor with invasion or adhesion of organs and structures, such as recurrent laryngeal nerve, esophagus, trachea, larynx, encirclement of neck large vessels, mediastinal vessels, extensive invasion of skin, subcutaneous soft tissue or neck muscles; 2). AJCC T4 Stage; 3). Difficult to achieve R0/R1 resection during preoperative assessment;
* Age 14-75 years;
* At least one measurable lesion (RECIST 1.1);
* Eastern Cooperative Oncology Group (ECOG) score 0-1;
* Expected survival time ≥ 12 weeks;
* The main organ functions meet the following criteria: Absolute neutrophil value (ANC) ≥ 1.5 × 109 / L; Platelet (PLT) ≥80 × 109 / L; Hemoglobin (HB) ≥9g / dL; White blood cell count> 1.5 × 109 / L; Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN, if with liver metastases, ALT and AST ≤ 5 ULN; Serum creatinine (Cr) ≤ 1.5 ULN or creatinine clearance (CCr) ≥ 50ml / min;
* Subjects of potential fertility are required to use at least one medically approved contraceptive method (such as an intrauterine device, contraceptive pill, or condom) during the study treatment and for 180 days after the end of the study treatment; The serum HCG test must be negative before the first medication.

Exclusion Criteria:

* Prior treatment with anti-angiogenic small molecule targeted drugs;
* Received other anti-tumor therapy (including but not limited to chemotherapy, radiotherapy, etc.) within 4 weeks prior to treatment, except for TSH suppression treatment;
* Allergy to the study drug ;
* Have a history of serious cardiovascular and cerebrovascular diseases;
* Patients whose imaging showed that the tumor had invaded the important blood vessels or the researchers judged that the tumor was likely to invade important blood vessels during the subsequent study period and caused fatal bleeding;
* Patients with hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
* The patient has had other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* The investigator considered that the subject was not suitable to participate in the study due to any clinical or laboratory abnormalities or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-04 (Estimated); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
ORR | approximately 1 years
  Objective Response Rate

SECONDARY OUTCOMES:
R0/1 resection rate | approximately 1 years
  R0 and R1 resection rate reviewed by operation team and pathologists R0 and R1 resection rate reviewed by operation team and pathologists R0 and R1 resection rate reviewed by operation team and pathologists dR0 and R1 resection rate reviewed by operation team and pathologists R0 and R1 resection rate reviewed by operation team and pathologists R0 and R1 resection rate reviewed by operation team and pathologists dvxddR0 and R1 resection rate reviewed by operation team and pathologists
DCR | approximately 1 years
  Disease Control Rate
PFS | approximately 1 years
  Progression Free Survival
AE | From first dose to within 30 days after the last dose
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jiaying Chen, Principal Investigator — Fudan University; Yu Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No